CLINICAL TRIAL: NCT05127447
Title: Effects of External Electric Stimulating in Individuals With Urinary Incontinence After Prostatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seyda TOPRAK CELENAY, associate professor, Ataturk Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/11/17
Record Dates: First submitted 2021-11-17; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Participants will be randomly divided into two groups (such as ES and sham groups)
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ES group (Experimental): External neuromuscular electrical stimulation was applied to the patients in supine position. It was applied for 30 minutes 3 days a week for 8 weeks. This stimulation consists of a total of eight external electrodes, including 2 sheaths wrapped around the thigh area and 4 electrodes for each leg. Electrodes were placed on the anterior and posterior proximal thighs, buttocks, and outside of the hips. The treatment protocol was applied with symmetrical biphasic current at a frequency of 50 Hertz (Hz), with stimulation and rest periods of 5 seconds of contraction and 5 seconds of rest.
  Interventions: Device: ES application
- Sham group (Sham Comparator): In the Sham group, for 45 minutes, 2 days a week, a vacuum electrode was connected from combined vacuum electrotherapy device over the pelvis and thigh, and only vacuum was applied while the patient was in the supine position, and no current was given from the applied device.
  Interventions: Other: Sham application

INTERVENTIONS:
Device: ES application — Electrical stimulation (ES) application will be given to the ES group
  Arms: ES group
Other: Sham application — Only vacuum was applied and no current was given from the applied device
  Arms: Sham group

SUMMARY:
The aim of this study is to investigate effects of external electric stimulating in individuals with urinary incontinence after prostatectomy.

DETAILED DESCRIPTION:
Urinary incontinence (UI) is common in men after prostotectomy, and patients' quality of life is adversely affected. In addition, electric stimulation (ES) can be played an important role in the management of UI . However, there are limitations in clearly demonstrating the effects of ES on men with UI after prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Being a male individual with stress or stress-dominant mixed UI symptoms after undergoing prostatectomy surgery for prostate cancer in the urology clinic
* Being over 40 years old
* Being 24 and over with Mini Mental Test results in individuals over 65 years of age.
* Not having residual cancerous tissue
* Volunteering to participate in the study

Exclusion Criteria:

* Having serious cardiovascular disease (unstable angina and arrhythmia patients, heart failure patients, etc.)
* Having sensory loss
* Having an ongoing urinary infection
* Having only urgency urinary incontinence
* Using a pacemaker
* Receiving active cancer treatment (radiotherapy, chemotherapy)
* Lack of evaluation parameters
* Not continuing the treatment regularly

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants with post-prostatectomy urinary incontinence
Enrollment: 40 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Pad Test | change from baseline at 8 weeks
  A 1-hour pad test will be applied. Beginning with an empty bladder, a pre-weighed sanitary napkin will be inserted into the underwear. The patient will be asked to drink 500 ml of water within 15 minutes and then remain active for half an hour. Then, various activities will be made to the patient to provoke involuntary urine leakage with a full bladder. weight will be measured.
UI symptoms | change from baseline at 8 weeks
  The ICIQ_SF is a UI questionnaire that evaluates symptom type and severity. It consists of 6 questions in total and the total score is 3., 4., 5. It is obtained by adding the scores they get from the questions

SECONDARY OUTCOMES:
Life quality | change from baseline at 8 weeks
  Life quality will be assessed with King's Health Questionnaire (KHQ).This questionnaire consists of two parts and 32 items.. The minimum possible score is 0 (best health) and the maximum possible score is 100 (worst health).
Sexual Function | change from baseline at 8 weeks
  Evaluation of sexual functions will be evaluated with International Index of Erectile Function IIEF-5 (IIEF-5), which is one of the most commonly used forms in men presenting with sexual complaints. It includes 5 main topics; erectile function, orgasm function, sexual desire, sexual intercourse satisfaction and general satisfaction are questioned with a total of 5 questions. Each question gets a score between 0-5. Total score; severe (5-7), moderate (8-11), mild-moderate (12-16), mild (17-21), no erectile dysfunction (22-25).
Evaluation of Subjective Improvement Perception | after treatment (8th week)
  The subjective improvement of UI symptoms pf the patients after treatment was evaluated using a 4-item Likert-type scale.
Evaluation of Treatment Satisfaction | after treatment (8th week)
  After the 8-week treatment program, the patients' satisfaction with the treatment for UI was evaluated using a 5-item Likert-type scale.

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Toprak Celenay, Principal Investigator — Ankara Yildirim Beyazıt University